CLINICAL TRIAL: NCT04556084
Title: Blinatumomab Bridging Therapy in High-Risk B-Acute Lymphoblastic Leukemia: A Phase 2 Study
Brief Title: Blinatumomab Bridging Therapy for BALL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Michael Burke (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Michael Burke, Associate Professor, Department of Pediatrics, Division of Hematology/Oncology/BMT, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Blina Part 1
Record Dates: First submitted 2020-09-09; First posted 2020-09-21 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; Refractory B Acute Lymphoblastic Leukemia; Relapsed B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Blinatumomab (Experimental): Up to 2 cycles of continuous infusion blinatumomab will be given based on the end of Cycle 1 disease response. Cycle 2 of blinatumomab can be given to subjects who have achieved remission (< 5% marrow blasts) after Cycle 1 but have persistent disease identified by multi-parameter flow cytometry (minimal residual disease (MRD) positive ≥ 0.01%) after Cycle 1.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab will be given as a 28-day continuous infusion with 14-days in between Cycle 1 and Cycle 2 as per the package insert and FDA approved labeling.
  Patient weight greater than or equal to 45kg will receive 28 mcg/day
  Patient weight less than 45kg will receive 15 mcg/m2/day
  Other Names: Blincyto

SUMMARY:
The investigator is testing the ability of a biologically active therapy in blinatumomab, an anti-CD19/CD3 bispecific T-cell engager, to further reduce residual leukemia immediately prior to HCT to improve post-HCT outcomes.

DETAILED DESCRIPTION:
The investigator is testing the ability of a biologically active therapy in blinatumomab, an anti-CD19/CD3 bispecific T-cell engager, to further reduce residual leukemia immediately prior to HCT to improve post-HCT outcomes. This Phase 2 study will determine the effectiveness of delivering 1 to 2 cycles of blinatumomab (Days 1-28) as bridging therapy in children, adolescent and young adults with relapse or persistent MRD B-ALL. Eligible subjects will receive 1 or 2, 28-day cycles of blinatumomab prior to proceeding to HCT. Centralized MRD assessment will be performed after completion of the 28-days of blinatumomab using both flow cytometry (University of Washington, Brent Wood, MD) and High-Throughput Deep Sequencing (HTS) MRD technologies (Adaptive Technologies, Seattle, WA). Subjects who achieve flow cytometry negative MRD (<0.01%) after a single cycle of blinatumomab can proceed directly to HCT whereas subjects who remain MRD positive by flow cytometry may receive a 2nd cycle of blinatumomab. Subjects who remain MRD positive by flow cytometry after a 2nd cycle of blinatumomab will come off study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B-ALL in hematologic complete remission (defined as an M1 marrow, < 5% blasts) with MRD in the bone marrow (≥ 0.01%) by multi-parameter flow cytometry and that meets one of the following:

  * Patients in first relapse or greater;

OR

• Patients with very-high risk biology ALL that is proceeding to HCT in first remission (e.g. Induction failure, Severe-hypodiploidy, Ph-like ALL);

OR

• Patients who have persistent MRD after Consolidation therapy (End of Consolidation (EOC) MRD positive ≥ 0.01%);

AND with the intent of going on to an allogeneic hematopoietic cell transplantation (HCT) independent of this study

* Patients must have an available donor and have intention of proceeding directly to HCT after completion of 1 to 2 cycles of Bridging therapy with blinatumomab.
* Age ≤ 25 years at time of study enrollment
* Karnofsky Performance Status ≥ 50% for patients 16 years and older and Lansky Play Score ≥ 50 for patients under 16 years of age (see Appendix 1)
* Have acceptable organ function as defined within 7 days of study registration:

Renal: creatinine clearance ≥ 60 mL/min/1.73m2 or serum creatinine based on age/gender

Hepatic: ALT < 5 x upper limit of normal (ULN) and total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age

Cardiac: left ventricular ejection fraction ≥ 40% by ECHO/MUGA

* At least 7 days must have elapsed from prior chemotherapy.
* Patients who have experienced their relapse after HCT are eligible, provided they have no evidence of acute or chronic Graft-versus-Host Disease (GVHD) and are off all transplant immune suppression therapy for at least 7-days (e.g. steroids, cyclosporine, tacrolimus). Steroid therapy for non-GVHD and/or non-leukemia therapy is acceptable.
* Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
* Monoclonal antibodies: At least 3 half-lives of the antibody must have elapsed after the last dose of monoclonal antibody (i.e. Inotuzumab = 12 days).
* Immunotherapy: At least 42 days after the completion of any type of immunotherapy (e.g. tumor vaccines or CAR T-cell therapy).
* XRT: Cranio or craniospinal XRT is prohibited during protocol therapy. ≥ 90 days must have elapsed if prior TBI, cranio or craniospinal XRT
* Sexually active females of child-bearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment and for 2 months after the last dose of chemotherapy. Sexually active men must agree to use barrier contraceptive for the duration of treatment and for 2 months after the last dose of chemotherapy.
* Voluntary written consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* History of CNS3 disease and/or active central nervous system (CNS) disease (≥ CNS2)
* Receiving concomitant chemotherapy, radiation therapy; immunotherapy or other anti-cancer therapy other than is specified in the protocol.
* Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Pregnant or lactating. The agents used in this study are known to be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. All females of childbearing potential must have a blood test or urine study within 7-days prior to the start of blinatumomab to rule out pregnancy.
* Known allergy to blinatumomab
* Participating in a concomitant Phase 1 or 2 study

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Burke, MD, Study Chair — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Blinatumomab: Up to 2 cycles of continuous infusion blinatumomab will be given based on the end of Cycle 1 disease response. Cycle 2 of blinatumomab can be given to subjects who have achieved remission (< 5% marrow blasts) after Cycle 1 but have persistent disease identified by multi-parameter flow cytometry (minimal residual disease (MRD) positive ≥ 0.01%) after Cycle 1.
  Blinatumomab: Blinatumomab will be given as a 28-day continuous infusion with 14-days in between Cycle 1 and Cycle 2 as per the package insert and FDA approved labeling.
  Patient weight greater than or equal to 45kg will receive 28 mcg/day
  Patient weight less than 45kg will receive 15 mcg/m2/day
Period: Overall Study
Arm/Group | Blinatumomab
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Blinatumomab
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 14 [9 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2
Peripheral White Blood Cell Count (from initial diagnosis) [Mean (Full Range); unit: 10*3 cells/mcL] | 4.7 [3 to 6.4]
CNS Status (from initial diagnosis) [Count of Participants; unit: Participants] — This baseline measure describes the CNS staging (from initial diagnosis) for the participants.
  CNS I - In cerebrospinal fluid (CSF) absence of blasts on cytospin preparation, regardless of number of white blood cells.
  CNS II - In CSF, cytospin positive for blasts in the presence of < 5/uL WBCs (or a traumatic LP) CNS III - In CSF, cytospin positive for blasts in the presence of >/=m 5/uL WBCs. Or signs of CNS leukemia.
  Participants
    CNS I | 2
    CNS II | 0
    CNS III | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects in Complete Remission (CR)
Description: The primary efficacy variable is the percent of subjects that remain in Complete Remission (CR) after completion of 1 or 2 cycles of blinatumomab. Complete remission was defined as <5% blasts in the bone marrow. Complete remission was further defined as minimal residual disease (MRD) positive (>/= to 0.01%) or MRD negative (<0.01%) as measured by flow cytometry of the bone marrow.
Time Frame: 1 or 2 Months depending on the number of cycles of blinatumomab
Measure: Number; unit: percentage of patients MRD negative
Arm/Group | Blinatumomab
Number analyzed (Participants) | 2
percentage of patients MRD negative | 100

2. Primary Outcome: Percentage of Subjects Flow Cytometry (FC) -Minimal Residual Disease (MRD) Negative Defined as <0.01% Leukemia
Description: The primary efficacy variable is the percent of subjects that become Flow Cytometry-MRD negative (FC-MRD negative) < 0.01% after completion of 1 or 2 cycles of blinatumomab.
Time Frame: 1 to 2 Months depending on the number of cycles of blinatumomab
Measure: Number; unit: percent of participants FC-MRD Negative
Arm/Group | Blinatumomab
Number analyzed (Participants) | 2
percent of participants FC-MRD Negative | 100

3. Secondary Outcome: Percentage of Subjects That Are High-Throughput Deep Sequencing (HTS)-Minimal Residual Disease (MRD) Negative Defined as Undetectable
Description: The percent of subjects that achieve MRD negative by molecular High-Throughput Deep Sequencing (HTS-MRD negative) (MRD undetectable) after completion of Blinatumomab bridging therapy, which may consist of 1 to 2 cycles of Blinatumomab.
Time Frame: After completion of Blinatumomab bridging therapy (1 participant's course consisted of 1 cycle, the other participant's course consisted of 2 cycles)
Measure: Number; unit: percentage of patients MRD negative
Arm/Group | Blinatumomab
Number analyzed (Participants) | 2
percentage of patients MRD negative | 100

ADVERSE EVENTS:
Time Frame: 4 weeks of treatment followed 4 weeks of follow-up
Description: AE does not differ from clinicaltrials.gov definitions
Arm/Group | Blinatumomab
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT04556084/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT04556084/ICF_001.pdf